CLINICAL TRIAL: NCT05325814
Title: Agreement Between Standard and Continuous Wireless Vital Sign Measurements Following Major Abdominal Surgery: A Clinical Comparison Study
Brief Title: Agreement Between Standard and Continuous Wireless Vital Sign Measurements
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Camilla Haahr-Raunkjaer, MD., Rigshospitalet, Denmark
Other Study IDs: WARD_SX_validation
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Patients
Keywords: wearable devices; continuous; comparison study; validation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Device: Continuous monitoring system: Continuous monitoring system Recruited patients will be continuously monitored with Isansys Lifetouch patch, Nonin WristOx 3150, Isansys wireless blood pressure monitor (Meditech Blue BP-05) and standard monitoring at the post anesthesia care unit

SUMMARY:
Patients undergoing major surgery are at risk of postoperative complications. Continuous wireless monitoring outside the post-anesthesia or intensive care units may enable early detection of patient deterioration, but good accuracy of measurements is required.

This validation study, which is part of the WARD-SX project, aimed to assess the agreement between vital signs recorded by standard and novel wireless devices

DETAILED DESCRIPTION:
Patients undergoing major surgery are at risk of postoperative complications. Complications may be preceded by abnormal vital signs. Standard monitoring at general wards is intermittent and manual, leaving the patients unobserved for extended periods.

The chance to enhance monitoring has arisen with recent technological advances in the form of small wearable and wireless devices that continuously record vital signs. Wearable devices enable continuous monitoring outside the intensive care unit and post-anesthesia care unit, thus enabling early detection of patient deterioration. However, before implementing such devices in hospital settings, good accuracy, and precision of measurements is required.

This validation study, which is part of the WARD-SX project, aimed to assess the agreement between vital signs recorded by standard and novel wireless devices

ELIGIBILITY:
Inclusion Criteria:

* ≥60 years, scheduled for major abdominal cancer surgery with planned PACU admission.

Estimated surgical intervention duration ≥2 hours.

Exclusion Criteria:

* Implanted cardioverter defibrillator or pacemaker, allergy to study devices, severe cognitive impairment assessed by Mini-Mental State Examination ≤24, or inability to cooperate in wearing the wireless monitoring equipment.

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planned for major abdominal surgery at Bispebjerg and Frederiksberg, and Rigshospitalet.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Heart rate comparisons | 1.5 hours (measurement interval every 15 min)
  Heart rate (beats per minute) measurements compared between Isansys Lifetouch and standard monitoring (Phillips IntelliVue). Analysed using Bland Altman (BA) analysis to measure mean diference and limits of agreement between to methods. The BA analysis is corrected for repeated measures within each subject.
Respiratory rate comparisons | 1.5 hours
  Respiratory rate (breaths per minute) measurements compared between Isansys Lifetouch and observed counted measurements. Analysed using Bland Altman (BA) analysis to measure mean difference and limits of agreement between to methods. The BA analysis is corrected for repeated measures within each subject.
SpO2 measurements comparisons wireless vs. standard | 1.5 hours (measurement interval every 15 min)
  SpO2 (percent) measurements compared between Nonin WristOx 3150 and standard monitoring. Analysed using Bland Altman (BA) analysis to measure mean difference and limits of agreement between to methods. The BA analysis is corrected for repeated measures within each subject.
SpO2 measurements comparisons wireless vs. invasive | 1.5 hours
  SpO2 (percent) measurements compared between Nonin WristOx 3150 and arterial arterial oxygen saturation. Analysed using Bland Altman (BA) analysis to measure mean difference and limits of agreement between to methods. The BA analysis is corrected for repeated measures within each subject.
Pulse rate comparisons | 1.5 hours
  Pulse rate measurements (beats per minute) measures compared between Nonin WristOx 3150 and standard monitoring. Analysed using Bland Altman (BA) analysis to measure mean difference and limits of agreement between to methods. The BA analysis is corrected for repeated measures within each subject.
Blood pressure comparisons wireless vs. standard | 1.5 hours, every 15 min
  Blood pressure (mmHg) measurements compared between Meditech BlueBp-05 and standard monitoring. Analysed using Bland Altman (BA) analysis to measure mean difference and limits of agreement between to methods. The BA analysis is corrected for repeated measures within each subject.
Blood pressure comparisons, wireless vs. arterial BP | 1.5 hours
  Systolic and diastolic (mmHg) measurements compared between Meditech BlueBp-05 and invasive arterial blood pressure. Analysed using Bland Altman (BA) analysis to measure mean difference and limits of agreement between to methods. The BA analysis is corrected for repeated measures within each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Eske K Aasvang, Dr. Med, Study Chair — Rigshospitalet, Denmark; Camilla Haahr-Raunkjaer, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Anesthesiology, Center for Cancer and Organ Diseases, Copenhagen, Denmark